CLINICAL TRIAL: NCT01646671
Title: A Multi-center, Open Label Study for Evaluation of the Safety, Tolerability and Efficacy of 8-week Treatment With LCZ696 in Japanese Patients With Severe Hypertension
Brief Title: Safety and Tolerability and Efficacy of LCZ696 in Japanese Severe Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696A1305
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Severe Hypertension
Keywords: Hypertension, Severe, LCZ696
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LCZ696 200 mg (Experimental): All participants were started on LCZ696 200 mg once daily on day 1. Participants who achieved mean sitting diastolic blood pressure (msDBP) of < 100 mmHg and mean sitting systolic blood pressure (msSBP) of < 160 mmHg at week 2 or a msDBP < 90 mmHg and msSBP < 140 mmHg at or after week 4 and for the duration of the study continued at 200 mg LCZ696 once daily.
  Interventions: Drug: LCZ696
- LCZ696 400 mg (Experimental): All participants were started on LCZ696 200 mg once daily on day 1. For participants who did not achieve mean sitting diastolic blood pressure (msDBP) of < 100 mmHg and mean sitting systolic blood pressure (msSBP) of < 160 mmHg at week 2 or a msDBP < 90 mmHg and msSBP < 140 mmHg at or after week 4, and did not have any signs of safety concerns, the LCZ696 dose was increased to 400 mg once daily.
  Interventions: Drug: LCZ696
- LCZ696 400 mg plus other hypertension (HTN) medications (Experimental): All participants were started on LCZ696 200 mg once daily on day 1. For participants who received LCZ696 400 mg and did not achieve msDBP < 90 mmHg and msSBP < 140 mmHg at or after week 4 and had no signs of safety concerns, another class of antihypertensive drugs (other than Angiotensin II receptor blockers or Angiotensin Converting Enzyme Inhibitor (ACEi) could be added, or the dose of concomitant antihypertensive drugs could be increased as per the package insert. Participants who received LCZ696 400 mg once daily did not change their dose for the remainder of the study.
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696 — LCZ696 200 mg tablet once daily
  Arms: LCZ696 200 mg
Drug: LCZ696 — 2 tablets of LCZ696 200 mg once daily titrated up from 1 tablet of 200 mg once daily
  Arms: LCZ696 400 mg
Drug: LCZ696 — 2 tablets of LCZ696 200 mg once daily titrated up from 1 tablet of 200 mg once daily plus other HTN medications
  Arms: LCZ696 400 mg plus other hypertension (HTN) medications

SUMMARY:
This study assessed the safety, tolerability, and efficacy of LCZ696 in severe hypertensive Japanese patients

DETAILED DESCRIPTION:
Summaries for treatment-emergent adverse events, serious adverse events and death were provided by the following actual treatment regimen (actual treatment patients received) in addition to all patients: LCZ696 200mg, 400mg, 400mg+other hypertensive medications.

Summaries for others than above were provided by the following treatment regimen (determined by the maximal treatment patients received) in addition to all patients: LCZ696 200mg, 400mg, 400mg+other hypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy office msSBP ≥180 mmHg or office msDBP ≥110 mmHg at baseline

Exclusion Criteria:

* Patients show msSBP ≥220 mmHg and/or msDBP ≥120 mmHg
* History of angioedema, drug-related or otherwise, as reported by the patient
* Patients unwilling or not able to discontinue safely the use of current antihypertensive medications during the study, as required by the protocol.
* Patients have significant cardiovascular co-morbidities
* Patients who previously entered a LCZ696 study and had been randomized or enrolled into the active drug treatment epoch.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Japan (8):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shibuya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo

REFERENCES:
- [Result] Kario K, Tamaki Y, Okino N, Gotou H, Zhu M, Zhang J. LCZ696, a First-in-Class Angiotensin Receptor-Neprilysin Inhibitor: The First Clinical Experience in Patients With Severe Hypertension. J Clin Hypertens (Greenwich). 2016 Apr;18(4):308-14. doi: 10.1111/jch.12667. Epub 2015 Sep 24. PMID 26402918

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications
Started | 3 | 11 | 21
Completed | 3 | 11 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treatment Assignment Set (TRTAG): This set included all patients who entered the treatment epoch.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications | Total
Number analyzed (Participants) | 3 | 11 | 21 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.0 (4.0) | 56.0 (12.24) | 49.3 (7.57) | 51.3 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2
  Male | 3 | 9 | 21 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events and Deaths
Description: Adverse events, serious adverse events deaths were monitored from screening to week 8.
Time Frame: Week 8
Population: AE analysis was determined by actual treatment, i.e. the LCZ696 dose and use of newly introduced anti-HTN medication/dose escalation of base anti-HTN medication on the day in which the corresponding summary was targeting. Participants could be counted in more than one category. Other safety analysis was determined by the maximum treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Total Participants: All participants who were treated
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications | Total Participants
Number analyzed (Participants) | 35 | 32 | 21 | 35
Percentage of participants
  Adverse Events (serious and non-serious) | 20.0 | 12.5 | 33.3 | 48.6
  Serious Adverse Events | 2.9 | 0 | 0 | 2.9
  Deaths | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in msSBP and msDBP at Week 8
Description: Sitting BP measurements were performed at screening through the end of study at every visit. Four separate sitting BP measurements were obtained with a full two-minute interval between measurements. The 4 measurements were summed and averaged, and then the baseline BP value was subtracted from the average value to get the change from baseline value.
Time Frame: Baseline, 8 weeks
Population: Full Analysis Set: included all patients who entered the treatment epoch. This set was determined by the maximum treatment patients received, i.e. combination of the highest LCZ696 dose and use of newly introduced anti-HTN medication/dose escalation of base anti-HTN medication during the treatment epoch.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications | Total Participants
Number analyzed (Participants) | 3 | 11 | 21 | 35
mmHg
  msSBP | -48.83 (11.730) | -30.34 (15.054) | -35.98 (15.229) | -35.31 (15.348)
  msDBP | -34.25 (7.378) | -16.98 (7.394) | -23.08 (8.514) | -22.12 (9.167)

3. Secondary Outcome: Percentage of Participants With Successful Blood Pressure (BP) Control in msSBP/msDBP at End of Study
Description: Successful BP control in patients with severe hypertension at the end of study treatment was defined as follows: msSBP/msDBP< 140/90 mmHg.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications | Total Participants
Number analyzed (Participants) | 3 | 11 | 21 | 35
Percentage of Participants | 66.7 | 18.2 | 47.6 | 40.0

4. Secondary Outcome: Percentage of Participants Achieving Successful msSBP Control at End of Study
Description: Successful msSBP control in patients with severe hypertension at the end of study treatment was defined as msSBP <140 mmHg.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications | Total Participants
Number analyzed (Participants) | 3 | 11 | 21 | 35
Percentage of Participants | 100 | 45.5 | 66.7 | 62.9

5. Secondary Outcome: Percentage of Participants Achieving Successful msDBP Control at End of Study
Description: Successful msDBP control in patients with severe hypertension at the end of study treatment was defined as msDBP < 90 mmHg.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications | Total Participants
Number analyzed (Participants) | 3 | 11 | 21 | 35
Percentage of Participants | 66.7 | 36.4 | 52.4 | 48.6

6. Secondary Outcome: Percentage of Participants With SBP Response at End of Study
Description: SBP response was defined as <140 mmHg or a reduction ≥ 20 mmHg from baseline.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications | Total Participants
Number analyzed (Participants) | 3 | 11 | 21 | 35
Percentage of Participants | 100 | 81.8 | 85.7 | 85.7

7. Secondary Outcome: Percentage of Participants With DBP Response at End of Study
Description: DBP response was defined as <90 mmHg or a reduction ≥ 10 mmHg from baseline.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg Plus Other Hypertension (HTN) Medications | Total Participants
Number analyzed (Participants) | 3 | 11 | 21 | 35
Percentage of Participants | 100 | 100 | 100 | 100

ADVERSE EVENTS:
Description: SAE and other AE analyses were determined by actual treatment, i.e. the LCZ696 dose and use of newly introduced anti-HTN medication/dose escalation of base anti-HTN medication on the day in which the corresponding summary was targeting. Participants could be counted in more than one category.
Groups:
- LCZ 200 mg: LCZ 200 mg
- LCZ 400 mg: LCZ 400 mg
- LCZ 400 mg + Other HTN Medications: LCZ 400 mg + other HTN medications
Arm/Group | LCZ 200 mg | LCZ 400 mg | LCZ 400 mg + Other HTN Medications | Total Participants
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/32 | 0/21 | 1/35
Other Adverse Events (participants affected / at risk) | 4/35 | 2/32 | 5/21 | 10/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ 200 mg (N=35) | LCZ 400 mg (N=32) | LCZ 400 mg + Other HTN Medications (N=21) | Total Participants (N=35)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ 200 mg (N=35) | LCZ 400 mg (N=32) | LCZ 400 mg + Other HTN Medications (N=21) | Total Participants (N=35)
NASOPHARYNGITIS (Infections and infestations) | 1 | 2 | 3 | 6
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 | 0 | 1 | 3
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.